CLINICAL TRIAL: NCT00432965
Title: KCI VAC Protocol VAC2001-08, "A Randomized, Controlled Multicenter Trial of Vacuum Assisted Closure Therapy™ in the Treatment and Blinded Evaluation of Diabetic Foot Ulcers"
Brief Title: Randomized, Controlled Multicenter Trial of Vacuum Assisted Closure Therapy™ in Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC2001-08
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcers
Keywords: Wound closure; Accelerated healing
MeSH Terms: conditions — Diabetic Foot

ARMS (2):
- VAC Therapy (Experimental): Treatment of Diabetic Foot Ulcers with VAC Therapy
  Interventions: Device: VAC Therapy
- Moist Wound Therapy (Active Comparator): Moist Wound Therapy (standard of care)
  Interventions: Device: Moist Wound Therapy

INTERVENTIONS:
Device: Moist Wound Therapy — Moist Wound Therapy (Standard of Care)
  Arms: Moist Wound Therapy
Device: VAC Therapy — VAC Therapy
  Other Names: NPWT
  Arms: VAC Therapy

SUMMARY:
To determine if topical negative pressure therapy delivered by the V.A.C.® device is clinically efficacious and cost effective in the treatment of diabetic foot ulcers.

The purpose of this study is to compare the effectiveness of V.A.C.® Therapy to moist wound therapy of diabetic foot ulcers. The primary objective is to determine the effect of V.A.C.® Therapy on the incidence of complete wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a calcaneal, dorsal or plantar diabetic foot ulcer ≥ 2 cm2 in area after debridement. (If more than one ulcer is present, all wounds will be treated using the same method, but only one ulcer will be studied.)
* DFU equivalent to Stage 2 or greater, as defined by Wagner's Scale system (See Appendix E)
* Evidence of adequate perfusion by one of the following on the affected extremity,(within the past 60 days):Dorsum transcutaneous oxygen test (TcPO2) with results of ≥30 mmHg, or ABIs with results of ≥0.7 and ≤1.2 and toe pressures with results of ≥30 mmHg, or Doppler arterial waveforms, which are triphasic or biphasic at the ankle in the affected leg.
* Age ≥ 18 years of age
* HbA1c ≤ 12% (collected within the last 90 days.)
* Evidence of adequate nutrition by one of the following:
* Lab results reflecting Pre-Albumin >16 mg/dl and Albumin level is >3 g/dl (during the seven days prior to the study period), or a nutritional consult will be done and with appropriate supplementation started. Proper documentation on CRFs is needed.

Exclusion Criteria:

* Patients with recognized active Charcot abnormalities of the foot, as evidence by clinical symptoms that interfere with either randomized treatment group
* Ulcers resulting from electrical, chemical, or radiation burns, or venous insufficiency
* Untreated infection or cellulites at site of target ulcer
* Presence of untreated osteomyelitis
* Collagen vascular disease
* Malignancy in the ulcer
* Presence of necrotic tissue
* Uncontrolled hyperglycemia
* Concomitant medications that include (washout period of 30 days for corticosteroids, immunosuppressive medications, or chemotherapy)
* Open amputations
* Prior V.A.C. therapy within 30 days.
* Current or prior normothermic (Warm-UP®) or HBO therapy within 30 days.
* Current or prior treatment with recombinant or autologous growth factor products within the past 30 days. (Examples: Regranex or Procuren)
* Current or prior treatment with skin or dermal substitutes and dressings (Examples: Apligraft, Dermagraft, or Integra) with living cells capable of producing growth factors (Example: Oasis) within the past 30 days.
* Current use of any enzymatic debridment agent (Example: Acuzyme /Panafil) during the active treatment phase of the study
* Pregnant or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2002-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Blume, DPM, Principal Investigator — North American Center for Limb Preservation
Locations (25):
- United States (24):
  - Maricopa Medical Center, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Tucson Vascular Surgery, PLLC, Tucson, Arizona
  - Southern Arizona VA Medical Center, Dept. Surgery, Tucson, Arizona
  - Bay Area Foot Care, Castro Valley, California
  - Innovative Medical Technologies, Los Angeles, California
  - Walter F. D Costa, Santa Rosa, California
  - Banner Health at North Colorado Med. Ctr, Greeley, Colorado
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Bay Pines VA Medical Center, Bay Pines, Florida
  - Podiatric Success, Inc., Boca Raton, Florida
  - Aim Research, Atlanta, Georgia
  - Hines VA Hospital, Hines, Illinois
  - North Chicago VAMC, North Chicago, Illinois
  - Rosalind Franklin University, North Chicago, Illinois
  - Des Moines University, Des Moines, Iowa
  - St. Lukes Roosevelt, New York, New York
  - East Carolina University, Greenville, North Carolina
  - Circleville Foot and Ankle, LLC, Circleville, Ohio
  - Genesis Health Care System, Zanesville, Ohio
  - Valley Baptist Medical Center, Brownsville, Texas
  - Robert Wunderlich, DPM, San Antonio, Texas
  - Abbott Clinical Research, Inc., San Antonio, Texas
  - Madigan Army Hospital, Tacoma, Washington
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VAC Therapy | Moist Wound Therapy
Started | 169 | 166
Completed | 75 | 80
Not Completed | 94 | 86
Not completed — Lost to Follow-up | 22 | 19
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Physician Decision | 14 | 13
Not completed — Lack of Efficacy | 8 | 13
Not completed — Non-compliance | 7 | 0
Not completed — Adverse Event | 22 | 19
Not completed — Death | 3 | 4
Not completed — Exclusionary Methods | 1 | 2
Not completed — Incomplete Data | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAC Therapy | Moist Wound Therapy | Total
Number analyzed (Participants) | 169 | 166 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.3) | 58.9 (11.51) | 58.1 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 44 | 72
  Male | 141 | 122 | 263
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 28 | 22 | 50
  Race/Ethnicity: Caucasian | 95 | 100 | 195
  Race/Ethnicity: Hispanic | 41 | 40 | 81
  Race/Ethnicity: Native American | 3 | 3 | 6
  Race/Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 4 | 4 | 8
  United States | 165 | 162 | 327

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Complete Ulcer Closure Closure.
Time Frame: Days 0-114
Population: Analysis of this endpoint was based on the Intent-to-Treat (ITT population). Subjects who signed an informed consent and were randomized, but failed to undergo their assigned randomized treatment, were included in this population.
Measure: Count of Participants; unit: Participants
Arm/Group | VAC Therapy | Moist Wound Therapy
Number analyzed (Participants) | 162 | 162
Participants
  Days 0-7 | 1 | 1
  Days 8-14 | 3 | 2
  Days 15-28 | 8 | 2
  Days 29-42 | 8 | 9
  Days 43-56 | 12 | 11
  Days 57-84 | 21 | 10
  Days 85-114 | 14 | 9
  Days 0-114 | 67 | 44
Statistical Analysis 1: Comparison: VAC Therapy vs Moist Wound Therapy; Time Frame: Days 0-114; Test type: Superiority; p = 0.007, Fisher Exact; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.19 to 3.02]

ADVERSE EVENTS:
Time Frame: Through Day 112; for those patients whose wound achieved ulcer closure they were followed through 9 months.
Arm/Group | VAC Therapy | Moist Wound Therapy
All-Cause Mortality (participants affected / at risk) | 4/169 | 5/166
Serious Adverse Events (participants affected / at risk) | 59/169 | 61/166
Other Adverse Events (participants affected / at risk) | 112/169 | 71/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAC Therapy (N=169) | Moist Wound Therapy (N=166)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 3
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 5
Cataract (Eye disorders) | 1 | 0
Eye Haemorrhage (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 2
Non-cardiac Chest Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 12 | 11
Osteomyelitis (Infections and infestations) | 9 | 16
Infected Skin Ulcer (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 3 | 2
Bacteraemia (Infections and infestations) | 2 | 0
Central Line Infection (Infections and infestations) | 2 | 1
Gangrene (Infections and infestations) | 2 | 5
Pneumonia (Infections and infestations) | 2 | 2
Staphylococcal Infection (Infections and infestations) | 2 | 2
Wound Infection (Infections and infestations) | 2 | 5
Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 1
Catheter Sepsis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 1 | 3
Staphylococcal Sepsis (Infections and infestations) | 1 | 1
Thrombophlebitis Septic (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Kidney Infection (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Graft Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Wound Decomposition (Injury, poisoning and procedural complications) | 1 | 0
Vascular Graft Complication (Injury, poisoning and procedural complications) | 0 | 2
Cardiac Enzymes Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 1
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 2
Renal Impairment (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0
Wound Debridement (Surgical and medical procedures) | 0 | 1
Femoral Artery Occlusion (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAC Therapy (N=169) | Moist Wound Therapy (N=166)
Oedema Peripheral (General disorders) | 9 | 10
Cellulitis (Infections and infestations) | 8 | 8
Wound Infection (Infections and infestations) | 16 | 10
Wound Complication (Injury, poisoning and procedural complications) | 19 | 10
Skin Maceration (Skin and subcutaneous tissue disorders) | 101 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days